CLINICAL TRIAL: NCT01883479
Title: Effect of Exercise and Wellness Interventions on Preventing Postpartum Depression.
Acronym: HM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH096748 (NIH); R01MH096748 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-06-21 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Exercise; Health; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Experimental): Telephone-based intervention designed to increase exercise among postpartum women.
  Interventions: Behavioral: Exercise
- Wellness/Support (Experimental): Telephone-based intervention designed to provide support to postpartum women.
  Interventions: Behavioral: Wellness/Support
- Usual care (No Intervention): Participants receive usual care and will receive their choice of the interventions at 9 months.

INTERVENTIONS:
Behavioral: Exercise — Telephone-based intervention designed to increase exercise among postpartum women.
  Arms: Exercise
Behavioral: Wellness/Support — Telephone-based intervention designed to provide support to postpartum women.
  Arms: Wellness/Support

SUMMARY:
The purpose of this study is to examine the efficacy of the active interventions (exercise or wellness/support intervention) compared to usual care on the prevention of postpartum depression among women at risk for depression. The investigators will also examine the efficacy of an exercise intervention compared to a wellness/support intervention on postpartum depressive symptoms among women at risk for depression.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of exercise and wellness/support interventions for preventing postpartum depression. Specifically, 450 sedentary postpartum women (2-6 weeks postpartum) with a history of depression prior to pregnancy will be randomized to one of three groups each lasting six months: (1) telephone-based exercise intervention; (2) telephone-based wellness/support intervention; or (3) usual care. Participants will also complete a follow-up assessment session at 9 months. Participants will be recruited via online, email, and print advertisements. The investigators will obtain healthcare provider consent for each participant prior to randomization. The exercise intervention will consist of a theory-based telephone intervention shown to increase exercise among postpartum women in a previous study (Lewis et al., 2011). The wellness/support condition will be on the same schedule as the exercise intervention and will address several topics related to wellness. The usual care condition will receive their choice of the exercise or wellness/support condition upon completion of their final assessment. The primary dependent variable will be depression as measured by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) and the Edinburgh Postnatal Depression Scale (EPDS). Exercise adherence will be assessed using the 7-Day Physical Activity Recall Interview and the ActiGraph (i.e., an accelerometer, an objective measure of exercise).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Low active
* Currently pregnant (who will wait to be randomized until postpartum) or less than six weeks postpartum
* History of depression

Exclusion Criteria:

* Less than 18 years of age
* Pre-existing hypertension or diabetes
* Currently exercising (defined as exercising more than 60 minutes per week)
* Enrolled in another exercise or weight management study
* Another member of the household participating in the study
* Unable to exercise for 20 minutes continuously
* Musculoskeletal problems such as arthritis, gout, osteoporosis, or back, hip or knee pain that may interfere with exercising
* Exercise induced asthma
* Any condition that would make exercise unsafe or unwise
* Taking medication that interferes with heart rate response to exercise such as beta blockers
* Hospitalization for a psychiatric disorder in the past six months
* Current depressive episode (based on the SCID) and/or currently receiving antidepressant medication or psychotherapy for depression (participants who are depressed prior to randomization will be referred to their primary physician or psychiatrist)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2012-12; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Depression | 6 months
  Depression assessed by the The Structured Clinical Interview for DSM-IV Axis I Disorders; SCID-I

SECONDARY OUTCOMES:
Depressive Symptoms | 6 months
  Depressive symptoms as assessed by the PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Lewis, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lewis BA, Schuver K, Dunsiger S, Samson L, Frayeh AL, Terrell CA, Ciccolo JT, Fischer J, Avery MD. Randomized trial examining the effect of exercise and wellness interventions on preventing postpartum depression and perceived stress. BMC Pregnancy Childbirth. 2021 Nov 22;21(1):785. doi: 10.1186/s12884-021-04257-8. PMID 34802425